CLINICAL TRIAL: NCT03739294
Title: Urine Concentrations of Vilanterol After Inhaled Administration of Vilanterol/Fluticasone Furoate: Defining a Urine Threshold and Decision Limit for Vilanterol in Doping Control Analysis
Brief Title: Urine Concentrations of Vilanterol After Inhaled Administration of Vilanterol/Fluticasone Furoate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Vibeke Backer, Professor, Dr.med, Bispebjerg Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: WADAVIL2018
Record Dates: First submitted 2018-11-09; First posted 2018-11-13 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — fluticasone furoate-vilanterol trifenatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- PILOT: 4 puffs once (Experimental): 4 puffs of Fluticasone Furoate/ Vilanterol Trifenatate 184/22 micrograms
  Interventions: Drug: Fluticasone Furoate/ Vilanterol Trifenatate
- PILOT: 4 puffs once a day for 7 days (Experimental): 4 puffs of Fluticasone Furoate/ Vilanterol Trifenatate 184/22 micrograms for 7 days
  Interventions: Drug: Fluticasone Furoate/ Vilanterol Trifenatate
- LARGE: 4 puffs once (Experimental): Supra-therapeutic inhalation of Fluticasone Furoate/ Vilanterol Trifenatate 184/22 micrograms (4 puffs) once
  Interventions: Drug: Fluticasone Furoate/ Vilanterol Trifenatate
- LARGE: 4 puffs once a day for 7 days (Experimental): Supra-therapeutic inhalation of Fluticasone Furoate/ Vilanterol Trifenatate 184/22 micrograms (4 puffs) daily for 7 days
  Interventions: Drug: Fluticasone Furoate/ Vilanterol Trifenatate
- LARGE: 1 puff once (Experimental): Therapeutic inhalation of Fluticasone Furoate/ Vilanterol Trifenatate 184/22 micrograms (1 puff) once
  Interventions: Drug: Fluticasone Furoate/ Vilanterol Trifenatate
- LARGE: 1 puff once a day for 7 days (Experimental): Therapeutic inhalation of Fluticasone Furoate/ Vilanterol Trifenatate 184/22 (1 puff) daily for 7 days
  Interventions: Drug: Fluticasone Furoate/ Vilanterol Trifenatate

INTERVENTIONS:
Drug: Fluticasone Furoate/ Vilanterol Trifenatate — Asthma inhalation medication
  Other Names: Relvar Ellipta 184/22 micrograms

SUMMARY:
Introduction: The prevalence of asthma and exercise-induced bronchoconstriction is high in the athletic population. In endurance sport, the prevalence has been reported to be as high as 30-50% compared to the general population prevalence of approximately 5-10% in Western countries. First-line treatment in asthma is reliever medication and inhaled corticosteroids (ICS). Therefore, β2-adrenoceptor agonists and ICS are commonly prescribed drugs to athletes. Although long-acting β2-agonists (LABA) are the most commonly used β2-agonists in asthma management, development of ultra-long acting β2-agonists (U-LABA) as vilanterol may change this. U-LABA has a long duration of action (24 hours) compared with LABA (12 hours). The accumulated number of inhalations per day for elite athletes may thus be reduced when prescribed with U-LABA as compared to LABA. Use of β2-agonists are restricted by the World Anti-Doping Agency (WADA). As of 2018, β2-agonists salbutamol, formoterol and salmeterol are allowed by inhalation in therapeutic doses, whereas other β2-agonists, such as terbutaline and vilanterol still require the athlete to obtain a therapeutic use exemption (TUE). To discriminate therapeutic use from supra-therapeutic misuse, WADA has established urinary thresholds and decision limits based on urine concentrations of salbutamol, salmeterol and formoterol. However, while data on urine concentrations of these three β2-agonists are well-described in studies that simulate sport-specific situations that are applicable for doping control, no such data exist for the novel U-LABA vilanterol. For instance, asthmatic athletes using β2-agonists usually inhale the drug before training or competition as prophylaxis for bronchoconstriction. Thus, studies are needed to investigate the urine concentrations of vilanterol after inhaled administration in set-ups that are applicable to doping control which this study aims to investigate.

Method: The study is divided in two phases. The first phase consists of a pharmacokinetic pilot trial (EXP1). Depending on the analytical outcome of the pilot study, the study proceeds into the second phase, which is a larger pharmacokinetic trial (EXP2). Both EXP1 and EXP 2 are open label studies.

EXP1: 6 healthy, well trained individuals are recruited to perform two trial days. First trial day consists of inhalation of the study drug in 4 times therapeutic dose followed by an exercise session. Before second trial day subjects inhales 4 times the therapeutic dose at home and on day 7 perform a training session. Urine and blood are collected in the following 72 hours both days.

EXP2: 20 healthy, well trained individuals are recruited to perform four trial days in the same way as EXP1. But here both normal use and four times normal dose is investigated.

DETAILED DESCRIPTION:
OBJECTIVES The main objective of the present study is to investigate urine concentrations of vilanterol and its metabolites (GSK932009 and GW630200) after single dose inhalation of Relvar® (22/184 mcg VI/FF) at therapeutic and supratherapeutic doses. A secondary objective is to investigate whether vilanterol and its metabolites (GSK932009 and GW630200) are present at higher concentrations in urine after seven days of daily inhalation of Relvar® at therapeutic and supratherapeutic doses.

Applicability The results from the study will help establish a urine threshold and decision limit for vilanterol on the WADA list of prohibited substances, thus lessening the administrative burdens associated with TUEs.

Study drug Study treatment in this study is refers to either therapeutic dosage of 22/184 micrograms of vilanterol/fluticasone furoate or four times therapeutic dosage of vilanterol/fluticasone furoate (88/736 micrograms, 4 puffs).

METHODS Study design The study is divided in two phases. The first phase consists of a pharmacokinetic pilot trial (EXP1). Depending on the analytical outcome of the pilot study, the study proceeds into the second phase which is a larger pharmacokinetic trial (EXP2).

Progression from the pilot phase (EXP1) of the study to the second phase (EXP2) of the study depends on a successful pilot phase (EXP1). Success will be concluded provided the pilot phase generates adequate urine concentration data for vilanterol and/or its metabolites (GSK932009, GW630200) with values above the assay limits of quantitation for at least 8 hours post dose. The pilot phase urine concentration data, together with plasma concentration data, will also be used to estimate the urinary concentrations of vilanterol and/or its metabolites at therapeutic and supratherapeutic under various conditions. These estimates will be used to determine whether progression to the second phase of the study is feasible and has a high probability of success in achieving its objectives.

Type of study The study is an open-label study. The study is classified as a Phase II study investigating pharmacokinetics Screening In EXP1 and EXP2, subjects are examined by a medical doctor and electrocardiography (ECG) is performed. Furthermore, subjects' lung function is measured with a spirometer and maximal oxygen consumption (VO2max) and performance are determined during an incremental bike ergometer test to exhaustion. Prior to the test, subjects warm up for 15 min. Subjects are told to keep a cadence of 80-100 rpm during the test. During the warm-up and incremental test, gas exchange is measured breath-by-breath.

After the VO2max-test, inhaler technique is practiced with a demonstrator device.

Pharmacokinetic trials

In EXP1, subjects meet at the laboratory for two trials:

Trial A1: Supra-therapeutic inhalation of Relvar® 22/184 (4 puffs) once Trial A2: Supra-therapeutic inhalation of Relvar® 22/184 (4 puffs) daily for 7 days

In EXP2, subjects meet at the laboratory for four trials:

Trial A1: Supra-therapeutic inhalation of Relvar® 22/184 (4 puffs) once Trial A2: Supra-therapeutic inhalation of Relvar® 22/184 (4 puffs) daily for 7 days Trial B1: Therapeutic inhalation of Relvar® 22/184 (1 puff) once Trial B2: Therapeutic inhalation of Relvar® 22/184 (1 puff) daily for 7 days

During each of the trials, subjects meet in the morning after an overnight fast. A urine sample is collected and subjects ingest a standardized meal and drink. One hour after the meal, study drug is administered during supervision and subjects start performing 60 min of exercise on a bike ergometer. Exercise is based on subjects' individual VO2max. To simulate the shifts in intensity during real-life competitive stages, the exercise protocol is performed at various shifting intensities, but still at a relative load of subjects' VO2max for inter-individual comparisons. Subjects are allowed to drink water during the exercise.

After exercise, subjects remain inactive for the rest of the trial. Three hours after administration of the study drug, subjects receive a standardized lunch and drink.

Urine is collected 0-1, 1-2, 2-4, 4-6, 6-8, 8-12, 12-16, 16-24, 24-36, 36-48 and 48-72 h following administration (corresponding to 0-71 h post exercise).

Venous blood samples are collected through a catheter in the antecubital vein ½, 1½, 3, 5, 7 and 10 h following administration.

Detailed instructions for urine and blood sample collection, processing, storage and transportation will be provided in the Study Procedures Manual) Concerning the Pilot study (EXP1) and the main study (EXP2): Between trials 1 and 2, subjects receive a Relvar® inhaler for six days of home use of 4 puffs per day, which will be monitored by staff via Skype or Facetime video call at the same time of the day as during trial 1. Twenty-four hours after the sixth day of home inhalation, subjects meet for trial 2. In EXP1 Trial A1 and Trial A2 is separated with minimum one week to ensure washout. In EXP2, Trial A1 and A2 and B1 and B2 are separated by at least 1 week to ensure washout.

End of trial The trial is finished when the last patient has been at the last visit. Pilot study (EXP1) is estimated to end at the end of 2018 and the large study is estimated to end at the end of 2019.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age between 18 and 39 years, both included at time of screening
* Ability to correctly use the inhaler device
* Active at least 5 h pr. week (defined as endurance exercise)
* VO2-max classified as high or very high (table 1)(Astrand, 1960) measured during an incremental test to exhaustion at the screening visit
* Male or non-pregnant female
* Females of childbearing potential has to use one or more of the following highly effective methods for contraception in order to be included:

  * Vasectomized partner
  * Bilateral tubal occlusion
  * Sexual abstinence
  * Intrauterine device
  * Hormonal contraception
* Females who are considered to have no childbearing potential are

  * Bilateral tubal ligation
  * Bilateral oophorectomy
  * Complete hysterectomy
  * Postmenopausal defined as 12 months with no menses without an alternative medical cause
* Non-smokers
* No daily use of prescribed medication

Exclusion Criteria:

* Diagnosis of heart, pulmonary (including asthma in Global initiative for asthma (GINA) 2-5), intestinal and renal diseases
* Allergy towards the active drug or any substances used in the drug
* Non-compliance with the protocol

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Vilanterol and its metabolites | 72 hours post drug administration
  Urine concentrations of vilanterol and its metabolites (GSK932009 and GW630200) 0-72 hours post drug administration.
Vilanterol and its metabolites | 0-10 hours post drug administration
  Blood concentrations of vilanterol and its metabolites (GSK932009 and GW630200) 0-10 hours post drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Backer, Physician, Principal Investigator — Respiratory Research Unit, Bispebjerg Hospital
Locations (1):
- Respiratory research unit, Bispebjerg University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided